CLINICAL TRIAL: NCT06525207
Title: New Diagnostic Tools in the Evaluation of the Posterior Compartment of the Women Pelvic Floor
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Elizabeth Barba, Head of Neurogastroenterology and Motility section, Gastroenterology department, Hospital Clinic of Barcelona
Other Study IDs: HCB/2024/0523
Record Dates: First submitted 2024-07-17; First posted 2024-07-29 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Anal Incontinence; Obstructive Defecation
Keywords: Impedance Planimetry; High Definition Anorectal Manometry
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Anal incontinence group: Women with anal incontinence and no symptoms of constipation
  Interventions: Device: Impedance Planimetry, High-definition anorectal manometry and Pelvic Floor Ultrasonography
- Obstructive defecation group: Women with constipation and predominant symptoms of obstructive defecation, without symptoms of anal incontinence
  Interventions: Device: Impedance Planimetry, High-definition anorectal manometry and Pelvic Floor Ultrasonography
- Healthy volunteer group: Women without any defecation disorders
  Interventions: Device: Impedance Planimetry, High-definition anorectal manometry and Pelvic Floor Ultrasonography

INTERVENTIONS:
Device: Impedance Planimetry, High-definition anorectal manometry and Pelvic Floor Ultrasonography — Global morpho-functional assessment of the anal sphincter complex using Impedance Planimetry, High-definition anorectal manometry and Pelvic Floor Ultrasonography

SUMMARY:
The goal of this observational study is to evaluate the pressure and distensibility index of the anal sphincter complex using high-definition anorectal manometry and the Impedance Planimetry system in women with fecal incontinence or constipation, as well as in a group of healthy volunteer women. The main questions it aims to answer are:

Assess the diagnostic accuracy of the Impedance Planimetry system compared to high-definition anorectal manometry (HD-ARM) in patients with anal incontinence and obstructive defecation.

Evaluate the diagnostic accuracy of three-dimensional reconstruction of the anal sphincter complex using HD-ARM to identify anal sphincter complex lesions compared to pelvic floor ultrasonography.

Determine the impact on the quality of life in women with anal incontinence and obstructive defecation based on the severity of symptoms assessed by validated scales

Participants will undergo the following tasks:

Undergo high-definition anorectal manometry and Impedance Planimetry testing.

Undergo pelvic floor ultrasonography to assess structural and functional aspects

Complete validated scales to assess symptoms and quality of life related to anal incontinence and obstructive defecation.

ELIGIBILITY:
Inclusion Criteria:

* Anal incontinence group: Women over 18 years old with predominantly fecal incontinence symptoms (St Mark > 6 points) and without constipation (KESS score < 10 points)
* Obstructive defecation group: Women over 18 years old with constipation symptoms and obstructive defecation (KESS score ≥ 10 points) and without fecal incontinence symptoms (St Mark < 1 point).
* Control group (healthy volunteers): Women over 18 years old without fecal incontinence (St Mark < 1 point) or constipation (KESS score < 10 points).

Exclusion Criteria:

* Anal incontinence and obstructive defecation groups: presence of anorectal tumors, ileo-anal/rectal anastomosis, previous anorectal surgeries (except primary repair of obstetric anal sphincter injury), anal stenosis, anal fistula, anal fissure, previous pelvic radiotherapy, use of opioids except loperamide, and history of inflammatory bowel disease (IBD).
* Control group (healthy volunteers): exclusion criteria are the same as for the patients groups and also include any volunteer with a history of systemic sclerosis, diabetes affecting target organs or insulin dependence, neurological conditions (stroke, multiple sclerosis, spinal cord injury, cauda equina syndrome, polyneuropathies), and history of pelvic floor disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women presenting symptoms of posterior compartment pelvic floor dysfunction (such as anal incontinence or obstructive defecation) referred for anorectal manometry evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Assess the diagnostic accuracy of the Impedance Planimetry system in patients with anal incontinence, obstructive defecation and healthy women. | Baseline
  Assess the diagnostic accuracy of the Impedance Planimetry system by distensibility index of anal sphincter complex evaluated by the Impedance Planimetry system in patients with anal incontinence, obstructive defecation and healthy women.
  Unit of Measure: Distensibility Index (mm^2/mmHg)
Assess the diagnostic accuracy of the High-definition anorectal manometry in patients with anal incontinence, obstructive defecation and healthy women. | Baseline
  Assess the diagnostic accuracy of the High-definition anorectal manometry in patients with anal incontinence, obstructive defecation and healthy women.
  Unit of Measure: Pressure (mmHg)

SECONDARY OUTCOMES:
Asses the diagnostic accuracy of the functional topographic images obtained from High-definition anorectal manometry. | Baseline
  Asses the diagnostic accuracy of sphincter disorders (descending perineum syndrome, rectal prolapse, intussusception and sphincter defects) using functional three-dimensional topographic images obtained from high-definition anorectal manometry compared with pelvic floor ultrasonography.
Determine the impact on the quality of life in women with anal incontinence using the SF-12 questionnaire, based on the severity of the symptoms (St. Mark's score) | Baseline
  Determine the impact on the quality of life in women with anal incontinence using the SF-12 questionnaire, based on the severity of the symptoms (St. Mark's score)
  Questionnaires:
  * Short form 12 health survey questionnaire (SF-12). Range from 0 to 100, with higher scores mean better quality of life.
  * St. Mark's incontinence score (St. Mark). Range from 0 to 24, with higher scores indicating worse symptom severity.
Determine the impact on the quality of life in women with obstructive defecation using the SF-12 questionnaire, based on the severity of the symptoms (KESS score) | Baseline
  Determine the impact on the quality of life in women with obstructive defecation using the SF-12 questionnaire, based on the severity of the symptoms (KESS score)
  Questionnaires:
  * Short form 12 health survey questionnaire (SF-12). Range from 0 to 100, with higher scores mean better quality of life.
  * Knowles-Eccersley-Scott-Symptom Constipation Score (KESS). Range from 0 to 39, with higher scores indicating worse symptom severity.
Determine the impact on the quality of life in women with anal incontinence using the FIQLS questionnaire, based on the severity of the symptoms (St. Mark's score) | Baseline
  Determine the impact on the quality of life in women with anal incontinence using the FIQLS questionnaire, based on the severity of the symptoms (St. Mark's score)
  Questionnaires:
  * Fecal Incontinence Quality of Life Scale (FIQLS). Range from 29 to 116, with lower indicating a worse quality of life.
  * St. Mark's incontinence score (St. Mark). Range from 0 to 24, with higher scores indicating worse symptom severity.
Determine the impact on the quality of life in women with obstructive defecation using the CVE-20 questionnaire, based on the severity of the symptoms (KESS score) | Baseline
  Determine the impact on the quality of life in women with obstructive defecation using the CVE-20 questionnaire, based on the severity of the symptoms (KESS score)
  Questionnaires:
  * Quality of life specific questionnaire for constipated patients (CV-20). Range from 0 to 80, with higher scores mean better quality of life.
  * Knowles-Eccersley-Scott-Symptom Constipation Score (KESS). Range from 0 to 39, with higher scores indicating worse symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic of Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rezaie A, Iriana S, Pimentel M, Murrell Z, Fleshner P, Zaghiyan K. Can three-dimensional high-resolution anorectal manometry detect anal sphincter defects in patients with faecal incontinence? Colorectal Dis. 2017 May;19(5):468-475. doi: 10.1111/codi.13530. PMID 27657739
- [Background] Vollebregt PF, Rasijeff AMP, Pares D, Grossi U, Carrington EV, Knowles CH, Scott SM. Functional anal canal length measurement using high-resolution anorectal manometry to investigate anal sphincter dysfunction in patients with fecal incontinence or constipation. Neurogastroenterol Motil. 2019 Mar;31(3):e13532. doi: 10.1111/nmo.13532. Epub 2019 Jan 13. PMID 30637863
- [Background] Benezech A, Behr M, Bouvier M, Grimaud JC, Vitton V. Three-dimensional high-resolution anorectal manometry: does it allow automated analysis of sphincter defects? Colorectal Dis. 2015 Oct;17(10):O202-7. doi: 10.1111/codi.13017. PMID 26046765
- [Background] Everist R, Burrell M, Mallitt KA, Parkin K, Patton V, Karantanis E. Postpartum anal incontinence in women with and without obstetric anal sphincter injuries. Int Urogynecol J. 2020 Nov;31(11):2269-2275. doi: 10.1007/s00192-020-04267-8. Epub 2020 Mar 10. PMID 32157322
- [Background] Taithongchai A, Thakar R, Sultan AH. Management of subsequent pregnancies following fourth-degree obstetric anal sphincter injuries (OASIS). Eur J Obstet Gynecol Reprod Biol. 2020 Jul;250:80-85. doi: 10.1016/j.ejogrb.2020.04.063. Epub 2020 May 4. PMID 32408091